CLINICAL TRIAL: NCT02569463
Title: Safety and Efficiency Study of Low-dose IL-2 Treatment in Macrophage Activation Syndrome
Brief Title: Low-dose IL-2 ( Interleukin-2) Treatment in Macrophage Activation Syndrome（MAS）
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL2-MAS
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Macrophage Activation Syndrome
MeSH Terms: conditions — Macrophage Activation Syndrome | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low-does rhIL-2 therapy (Experimental): Recombinant Human Interleukin-2 (RhIL-2) was administered subcutaneously at a dose of 1 million IU every other day for 4 weeks
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Recombinant Human Interleukin-2 (RhIL-2) was administered subcutaneously at a dose of 1 million IU every other day for 4 weeks.
  Other Names: Recombinant Human Interleukin-2

SUMMARY:
The investigators evaluate the effectiveness and safeness of low-dose Recombinant Human Interleukin-2 （rhIL-2） for MAS.

DETAILED DESCRIPTION:
Autoimmune-associated macrophage activation syndrome (MAS), also known as secondary hemophagocytic lymphohistiocytosis (HLH), is a rapidly progressing life-threatening disease. VP16 (Etoposide) is a well-known standard therapy, but is associated with substantial adverse effects, especially myelosuppression and infections , while steroids and ciclosporin (CSA) are not always efficient in this disease.

The investigators hypothesized that low- dose IL-2 could be a novel therapy in MAS. This clinical study will test the efficacy and safety of low dose IL-2 treatment in MAS. The investigators perform a single-centre pilot trial with rhIL-2 in MAS. The investigators evaluate the effectiveness and safeness of low-dose IL-2 for MAS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Macrophage Activation Syndrome（MAS）
* MAS secondary to autoimmune disease, such as Adult onset still's disease (AOSD), juvenile rheumatoid arthritis (JRA) or Systemic Lupus Erythematosus (SLE).

Exclusion Criteria:

* Primary MAS
* Secondary to neoplasia, lymphoma and virus infection
* pre-treatment with Cyclosporine A
* relevant cardiac, pulmonary, neurologic or psychiatric disease
* life-Vaccination within 4 weeks before begin with study medication
* pregnant or breast-feeding
* weight under 45kg or more than 80kg

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Disease activity on the HScore (a Score for the Diagnosis of Reactive Hemophagocytic Syndrome) | 1month
  Examination of the therapeutic effects (improvement in HScore) of low dose IL-2 in patients with MAS

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Department of Rheumatology and Immunology,Peking University People's Hospital
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China